CLINICAL TRIAL: NCT01175863
Title: Fractional Flow Reserve- And Intra-vascular Ultrasound-Guided Percutaneous Coronary Intervention With Drug-Eluting Stents in Intermediate Coronary Artery Lesion (FAVOR Study)
Brief Title: Fractional Flow Reserve (FFR) Versus Intravascular Ultrasound (IVUS) in Intermediate Coronary Artery Disease
Acronym: FAVOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Seung-Jea Tahk, MD, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAVOR
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Stenosis
Keywords: intravascular ultrasound; fractional flow reserve
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravascular ultrasound (Active Comparator)
  Interventions: Device: Grey scale intravascular ultrasound (Galaxy or Virtual histology-Intravascular Ultrasound)
- Fractional flow reserve (Active Comparator)
  Interventions: Device: Pressure wire(Radi Medical Systems)

INTERVENTIONS:
Device: Grey scale intravascular ultrasound (Galaxy or Virtual histology-Intravascular Ultrasound) — minimal lumen area on Intravascular ultrasound
  Other Names: Galaxy (Boston Scientific); Virtual histology (Volcano)
  Arms: Intravascular ultrasound
Device: Pressure wire(Radi Medical Systems) — Fractional flow reserve measured by pressure wire
  Other Names: Pressure wire (Radi Medical Systems)
  Arms: Fractional flow reserve

SUMMARY:
This study is a prospective, randomized, multi-center, open label trial to compare the clinical outcomes and effectiveness of Intravascular ultrasound (IVUS) versus Fractional Flow Reserve (FFR) guided Percutaneous coronary intervention (PCI) with intermediate coronary artery lesion.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, open label, two arm designed multi-center trial. When diagnostic coronary angiogram shows that the target lesion is intermediate stenosis, IVUS and/or FFR will be performed in order to decide PCI or defer by 1:1 randomization. The patients would be followed up to 2 years clinically.

ELIGIBILITY:
Inclusion Criteria:

Clinical indication:

* Patients with angina or patients with documented silent ischemia
* Patients who are eligible for intracoronary stenting
* Age > 18 years old, < 75 years old

Angiographic indication:

* Intermediate coronary artery disease (30-70% diameter stenosis) by visual estimation
* Reference vessel diameter ≥ 3.0mm by visual estimation

Exclusion Criteria:

* Acute or old myocardial infarction
* Previous coronary artery bypass graft
* Left main disease (≥ 50% stenosis)
* In-stent restenosis lesion
* Chronic total occlusion
* Low ejection fraction (< 40 %)
* Graft vessel lesion
* History of bleeding diathesis or coagulopathy
* Limited life-expectancy (less than 1 year) due to combined serious disease
* Contra-indication to heparin, everolimus
* Contraindication to aspirin, clopidogrel or cilostazol
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (composite of cardiac death, myocardial infarction and target vessel revascularization) | 1 year

SECONDARY OUTCOMES:
Cardiac death | 1 and 2 years
Myocardial infarction (MI) | 1 and 2 years
Composite of cardiac death or myocardial infarction | 1 and 2 years
Target vessel revascularization (ischemia- and clinically-driven) | 1 and 2 years
Target lesion revascularization (ischemia- and clinically-driven) | 1 and 2 years
Stent thrombosis (Academic Research Consortium criteria) | 1 and 2 years
In-stent and in-segment late loss on angiographic follow-up | 1 year
In-stent and in-segment restenosis rate | 1 year
Incidence and angiographic pattern of restenosis | 1 year
Canadian Cardiovascular Society Classification status | 1 and 2 years
The number of anti-angina medication | 1 and 2 years
Incidence of percutaneous coronary intervention at intravascular ultrasound and fractional flow reserve-guided group | Baseline (day 0)
Major adverse cardiac events (composite of cardiac death, myocardial infarction and target vessel revascularization) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sejung-Jea Tahk, MD, PhD, Principal Investigator — Ajou University Medical Center, Ajou University School of Medicine
Locations (8):
- South Korea (8):
  - Keimyung university Dongsan medical center, Daegu
  - Inje University, Ilsan
  - Korea University Guro Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul national university hospital, Seoul
  - Yensei University Gangnam Severance Hospital, Seoul
  - Ajou University Medical Center, Suwon
  - Yeonsei Univeristy Wonju College of Medicine Wonju Christion Hospital, Wŏnju